CLINICAL TRIAL: NCT04221009
Title: Improving Sleep Apnea Treatment Adherence After Brain Injury: A Feasibility Study
Brief Title: Feasibility of Improving Sleep Apnea Treatment Adherence After Brain Injury
Acronym: FISATABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N3303-P
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-03

CONDITIONS: Sleep Apnea, Obstructive; Brain Injuries, Traumatic
Keywords: Feasibility Studies; Continuous Positive Airway Pressure; Psychotherapy, Brief; Cognitive Behavioral Therapy; Motivational Interviewing; Sleep Apnea, Obstructive; Brain Injuries, Traumatic; Veterans
MeSH Terms: conditions — Sleep Apnea, Obstructive; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be asked to participate in four treatment sessions. The 4-session intervention is derived from evidence-based Motivational Interviewing and Cognitive Behavior Therapy. Participants will complete study measures pre- and post-intervention. Then, they will participate in a post-intervention interview to gather information of acceptability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (single arm) (Experimental): This is a 4-session intervention derived from Motivational Interviewing and Cognitive Behavior Therapy and adapted with cognitive accommodations.
  Interventions: Behavioral: MI and CBT 4-session manualized intervention

INTERVENTIONS:
Behavioral: MI and CBT 4-session manualized intervention — This is a 4-session intervention derived from Motivational Interviewing and Cognitive Behavior Therapy and adapted with cognitive accommodations.

SUMMARY:
Background: Obstructive sleep apnea (OSA) is a sleep disorder common among Veterans with moderate-to-severe traumatic brain injury (TBI). Untreated OSA increases risk of poor health outcomes including cognitive impairment, declining mental and physical health, and premature mortality. Positive airway pressure (PAP) is the frontline treatment for OSA that effectively reduces many negative health consequences of the disease. Unfortunately, PAP adherence is poor. A recent study showed that 68% of Veterans with moderate-to-severe TBI and OSA were nonadherent to PAP therapy. Psychoeducation is the standard of care for OSA treatment with PAP, but on its own is insufficient for improving adherence. Alternatives to the standard of care include evidence-based behavioral interventions such as Motivational Interviewing (MI) and Cognitive-Behavioral Therapy (CBT) which have been shown to improve PAP adherence in general sleep clinic samples. Unfortunately, these evidence-based interventions (designed for cognitively intact individuals) have not been adapted to address PAP adherence in persons with moderate-to-severe TBI, who often require cognitive accommodations. The goal of this study is to test the feasibility of a novel manualized intervention, designed with cognitive accommodations, and informed by MI and CBT, to address PAP adherence in Veterans with TBI and OSA.

Study Aims: Study Aim 1 tested the feasibility and acceptability of delivering the PAP adherence intervention. Study Aim 2 evaluated the feasibility of outcome and process measures.

Method: Veterans were recruited from inpatient and outpatient TBI and sleep clinics. Those meeting eligibility criteria (diagnosis of OSA and moderate-to-severe TBI; nonadherent to PAP, able to provide informed consent) were invited to participate in the 4-session intervention followed by a qualitative interview to inquire about intervention acceptability. Study measures (e.g., symptom severity, sleep quality of life), will be administered pre- and post-intervention.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is condition. The frontline treatment is Positive Airway Pressure (PAP) therapy. Adherence to PAP is essential to reap the therapeutic benefit of the treatment. Psychoeducation is part of the standard of care for the treatment of OSA, but on its own has been shown to be ineffective in improving PAP adherence. In persons without brain injury, alternatives to standard education, such as Motivational Interviewing (MI) and Cognitive Behavioral Therapy (CBT), have been shown to improve PAP adherence. To date, no published studies have examined maximizing frontline PAP treatment for persons with brain injury. Therefore, the objective of this study is to develop and test the feasibility of a manualized intervention, derived from evidence-based MI and CBT, and adapted with cognitive accommodations, to maximize PAP success in Veterans with OSA and TBI-related burden.

This is a 2-year mixed methods study using quantitative and qualitative inquiry to determine the feasibility and acceptability of a novel 4-session PAP adherence intervention (Aim 1). Feasibility is the ease to which the intervention can be delivered (e.g., eligibility rates, recruitment rates), and acceptability is the extent to which persons receiving the intervention consider it appropriate (e.g., satisfaction ratings). Feasibility of process and the ultimate outcome measures (e.g., completeness, perceived value and burden) will also be examined (Aim 2).

Participants will be recruited from clinics within the James A. Haley Veterans' Hospital (JAHVH), a tertiary care facility and teaching hospital. Participants will be recruited from three clinical settings: (1) inpatient TBI neurorehabilitation; (2) outpatient TBI clinics; and (3) sleep medicine clinic. Inclusion criteria for this study are as follows: (1) moderate-to-severe TBI; (2) diagnosed with OSA and prescribed PAP therapy; (3) are nonadherent to PAP treatment; and (4) able to consent. The plan is to enroll 19 participants, because -- using a conservative 75% retention estimate - it is expected that 14 will complete the intervention, exceeding the minimum for data saturation.

Upon receipt of consent, the pre-intervention study measures will be administered. Veterans will be scheduled for four treatment sessions. After the final session, participants will complete post-intervention measures. The intervention will be delivered by a doctoral level psychologist. Two independent evaluators will listen to 20% of audio-recorded sessions and conduct intervention fidelity checks using a Fidelity Rating Checklist created for this study by the PI, and adapted from other rating MI and CBT fidelity forms. Of the recordings, 10% will be the same session to conduct interrater reliability checks of the ratings. Participants will be contacted within 15 business days of their last intervention session for the qualitative interview to gather information on acceptability of the intervention. The project manager/research assistant will download objective PAP adherence data from the PAP software program during study pre-screening and 30 days following the last intervention session, to permit evaluation of adherence.

Analysis will include examination of persons enrolled and retained versus study eligible, and reasons for non-enrollment. Attendance will be described. Acceptability will be examined via the post-intervention interview. Identification of themes will be generated from the analysis using a constant comparative approach. The qualitative team will independently read the data, assign labels and codes to data segments, and develop initial themes, then meet to develop consensus on initial themes and codes, revising them using an iterative process, confirming evidence and consider rival explanations that contrast with findings and conclusions. Study measures. Pre- and post-intervention measures which will be examined for completeness. Descriptive data will be presented (e.g., central tendency, variability, change scores, and effect sizes).

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe TBI consistent
* diagnosed with OSA and prescribed PAP therapy
* nonadherent to PAP treatment
* are able to consent.

Exclusion Criteria:

* mild only TBI
* no TBI
* no OSA
* not prescribed PAP therapy
* adherent to PAP therapy (6) unable to provide consent on own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Silva, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Supporting Information: Study Protocol, ICF
Time Frame: Will be available starting twelve months following publication of study findings.
Access Criteria: Data are not publicly available. Information will be shared by contacting the study PI and upon institutional approval.

REFERENCES:
- [Derived] Silva MA, Arriola NB, Radwan CK, Womble BM, Healey EA, Lee JM, Aloia MS, Nakase-Richardson R. Improving sleep apnea treatment adherence after traumatic brain injury: A nonrandomized feasibility study. Rehabil Psychol. 2022 Nov;67(4):461-473. doi: 10.1037/rep0000473. PMID 36355639
- Available data/document: Informed Consent Form — https://arc.research.usf.edu/Prod/sd/Doc/0/DDRU7K2KMHLK9ECT12FPTMA60B/3S78A88933BKN7869JO1NSMT62.pdf
- Available data/document: Study Protocol — https://arc.research.usf.edu/Prod/sd/Doc/0/06USV5NTK2VKJ06CUK3TQJR578/Protocol%20v01%202019-10-24.docx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from inpatient TBI units and outpatient TBI clinics per IRB-approved protocol. The recruitment period occurred between August 2020 and December 2021.
Pre-assignment Details: All 17 participants who agreed to participate were enrolled in the study and assigned to the single arm of the study.
Groups:
- Intervention (Single Arm): This is a 4-session intervention derived from Motivational Interviewing and Cognitive Behavior Therapy and adapted with cognitive accommodations. MI and CBT 4-session manualized intervention: This is a 4-session intervention derived from Motivational Interviewing and Cognitive Behavior Therapy and adapted with cognitive accommodations.
Period: Overall Study
Arm/Group | Intervention (Single Arm)
Started | 17
Completed | 13 (4 participants were withdrawn from the study after enrollment because: no longer interested in participating (n=1), redeployed overseas thus no longer available (n=1), returned to full time employment and no longer interested (n=1) and ongoing computer technological problems precluding participation (n=1).)
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: Events per hour] | 22.9 (28.2)
Oxygenation Nadir [Mean (Standard Deviation); unit: % peripheral oxygen saturation] — Oxygen nadir during polysomnographic study measured via pulse oximeter was abstracted from existing medical records, per study protocol. Oxygen nadir is a metric that refers to the lowest point of peripheral oxygen saturation, which can range theoretically from 0% to 100%.
  % peripheral oxygen saturation | 86.0 (3.8)
Glasgow Outcome Scale-Extended (GOS-E) [Mean (Standard Deviation); unit: units on a scale] — The GOS-E is rated on an ordinal scale, 8 levels, ranging from 1 to 8 with higher scores indicating greater (better) outcome.
  units on a scale | 5.2 (1.4)
Fatigue Severity Scale (FSS) [Mean (Standard Deviation); unit: units on a scale] — The FSS is a 9-item measure of self-reported fatigue severity. Items are rated from 1 (disagree) to 7 (agree) with higher scores denoting greater symptom severity. Total scores range from 9 to 63. Higher scores reflect greater self-reported fatigue. Population: 1 participant did not complete the FSS
  units on a scale
    number analyzed (Participants) | 16
    (all) | 41.7 (15.2)
Functional Outcome of Sleep Questionnaire (FOSQ) [Mean (Standard Deviation); unit: units on a scale] — The FOSQ is a 30-item instrument. Each item is rated on a score from 1 to 4, with lower scores denoting worse functional impact (worse outcome). The 30 items represent functioning across 5 life domains. The 5 life domain scores are the average of the items within that domain. The total score (reported in this study) ranges from 5 to 20 and is an average of the 5 domain scores. Population: 2 participants did not complete the FOSQ
  units on a scale
    number analyzed (Participants) | 15
    (all) | 14.0 (4.1)
OSA Treatment Barriers Questionnaire (OTBQ) [Mean (Standard Deviation); unit: units on a scale] — The OTBQ is a 6-item self-report measure of perceived treatment barriers. Each item is rated on a score from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 6 to 30. Higher scores denoting greater perceived OSA treatment barriers. Population: 2 participants did not complete the OTBQ
  units on a scale
    number analyzed (Participants) | 15
    (all) | 13.3 (4.1)
Self Efficacy Measure for Sleep Apnea (SEMSA) Risk Perception [Mean (Standard Deviation); unit: units on a scale] — The SEMSA is a 26 item self-report measure of a person's perception of personal risk of susceptibility and consequences of untreated OSA (Risk Perception), expectations of personal health outcome following treatment for OSA (Treatment Outcome Expectancies), and perception that one can successfully manage their OSA (Self Efficacy). Each item is rated on a scale from 1 to 4.
  The SEMSA Risk Perception subscale is 8 items. Score range is 1 to 32, with higher scores denoting greater perceived risk. Population: 2 participants did not complete the SEMSA Risk Perception
  units on a scale
    number analyzed (Participants) | 15
    (all) | 15.9 (4.7)
Self Efficacy Measure for Sleep Apnea (SEMSA) Outcome Expectancies [Mean (Standard Deviation); unit: units on a scale] — The SEMSA is a 26 item self-report measure of a person's perception of personal risk of susceptibility and consequences of untreated OSA (Risk Perception), expectations of personal health outcome following treatment for OSA (Treatment Outcome Expectancies), and perception that one can successfully manage their OSA (Self Efficacy). Each item is rated on a scale from 1 to 4.
  The Treatment Outcome Expectancies subscale is 9 items. Score range is 1 to 36, with higher scores denoting greater perceived treatment benefit. Population: 2 participants did not complete the SEMSA Outcome Expectancies
  units on a scale
    number analyzed (Participants) | 15
    (all) | 28.2 (4.2)
Self Efficacy Measure for Sleep Apnea (SEMSA) Treatment Self-efficacy [Mean (Standard Deviation); unit: units on a scale] — The SEMSA is a 26 item self-report measure of a person's perception of personal risk of susceptibility and consequences of untreated OSA (Risk Perception), expectations of personal health outcome following treatment for OSA (Treatment Outcome Expectancies), and perception that one can successfully manage their OSA (Self Efficacy). Each item is rated on a scale from 1 to 4.
  The Self Efficacy subscale is 9 items. Score range is 1 to 36, with higher scores denoting greater perceived ability to manage their OSA. Population: 2 participants did not complete the SEMSA Treatment Self-Efficacy
  units on a scale
    number analyzed (Participants) | 15
    (all) | 23.7 (7.1)
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — The ESS is an 8-item measure. Items are rated from 0 to 4, with higher scores denoting greater symptom severity. Population: 2 participants did not complete the ESS
  units on a scale
    number analyzed (Participants) | 15
    (all) | 11.9 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Narrative Evaluation of Intervention Interview (Post-intervention Qualitative Interview)
Description: The Narrative Evaluation of Intervention Interview is a 16-item semi-structured interview that elicits participant feedback about an intervention. The data yielded by the NEII are qualitative, using qualitative thematic analysis. All 13 participants who completed the study also completed the NEII interview.
Time Frame: Post-intervention (up to 8 weeks after completion of the single arm intervention)
Measure: Number; unit: Themes
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 13
Themes | 4

2. Secondary Outcome: Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale is an 8-item validated measure of daytime sleepiness. Respondents rate how likely they are to doze in eight situations, each on a scale from 0 to 3. Scores range from 0 to 24. Higher scores representing greater levels of excessive sleepiness
Time Frame: Single time point, following completion of the single arm intervention, up to 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 13
units on a scale | 11.0 (5.0)

3. Secondary Outcome: Fatigue Severity Scale
Description: The Fatigue Severity Scale is a 9-item measure that is sensitive to change following OSA treatment. Respondents rate (on a scale from 1 to 7) the degree of fatigue symptoms experienced within the past 7 days. Total scores range from 9 to 63. Higher scores denote worse fatigue.
Time Frame: Single time point, following completion of the single arm intervention, up to 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 13
units on a scale | 36.4 (15.6)

4. Secondary Outcome: Functional Outcomes of Sleep Questionnaire
Description: The Functional Outcomes of Sleep Questionnaire is a 30-item instrument that measures the impact of excessive sleepiness on quality of life in five domains. Items are rated from 1 to 4. Scores range from 1 to 120. Lower scores denote greater impact on quality of life.
Time Frame: Single time point, following completion of the single arm intervention, up to 12 weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 13
units on a scale | 14.7 (3.7)

ADVERSE EVENTS:
Time Frame: Adverse events time frame was between August 2020 (starting enrollment) until June 2022 (end of study). For each participant, adverse events monitoring occurred between time of study enrollment and either (1) time completed all study procedures, or (2) time participant withdrew from study. The adverse event monitoring period lasted for 1 year and 10 months. For the study sample as a whole, the average monitoring period was 139.6 days (or an average of 20 weeks or 4.6 months).
Description: Definitions of adverse and serious adverse events are the clinicaltrials.gov definitions.
Arm/Group | Intervention (Single Arm)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04221009/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT04221009/SAP_002.pdf
  • Informed Consent Form (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT04221009/ICF_001.pdf